CLINICAL TRIAL: NCT03776435
Title: Carcinogenic Risk of CT in Patients With Appendicitis
Brief Title: CT Carcinogenic Risk in Patients With Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Ji Hoon Park, Associated Professor, Seoul National University Bundang Hospital
Other Study IDs: AppyCTcancer
Record Dates: First submitted 2018-12-13; First posted 2018-12-14 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Computed Tomography; Carcinogenesis; Radiation Exposure; Appendicitis
MeSH Terms: conditions — Carcinogenesis; Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CT-exposed group
  Interventions: Radiation: Abdomen CT
- CT-unexposed group
  Interventions: Radiation: Abdomen CT

INTERVENTIONS:
Radiation: Abdomen CT — Patients are divided into CT-exposed or unexposed group according to the presence of claims codes of abdominopelvic CT conducted within seven days before and after appendectomy. The seven-day threshold is arbitrarily determined considering the delay in the diagnosis of appendicitis and the postoperative examination for surgical complication.

SUMMARY:
The purpose of this study is to compare the incidence rate of leukemia between CT-exposed and CT-unexposed group in patients who underwent appendectomy in South Korea.

DETAILED DESCRIPTION:
South Korea has a single-payer healthcare system, administered by National Health Insurance Service (NHIS). As healthcare providers in South Korea need to claim reimbursement to NHIS for the vast majority of diagnostic and therapeutic procedures, the NHIS database enabled us to construct a large cohort who did or did not undergo CT for appendicitis. The purpose of this study is to compare the incidence rate of cancer between CT-exposed and CT-unexposed group in patients who underwent appendectomy in South Korea.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be entered in the cohort on the date of appendectomy under the diagnosis of appendicitis

Exclusion Criteria:

* (a) patients who had a cancer diagnosis before the date of appendectomy,
* (b) those who had prior experience of CT examination more than 7 days before appendectomy,
* (c) those who had syndromes or diseases predisposing cancers,
* (d) those whose diagnosis was changed to appendiceal cancer and
* (e) those whose follow-up duration was shorter than a lag period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent appendectomy under the diagnosis of appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
Age and sex-standardized incidence rate ratio (IRR) for malignancies of hematologic system | Cancer occurrence after a lag period (2 years)
  Hematologic malignancies are categorized into lymphomas, multiple myeloma, leukemias, myelodysplasia and others using ICD-10 codes.

SECONDARY OUTCOMES:
Age and sex-standardized incidence rate ratio (IRR) for malignancies of abdominal organs | Cancer occurrence after a lag period (2 years)
  age and sex-standardized IRRs for malignancies of abdominal organs for CT-exposed versus unexposed patients.
Age and sex-standardized incidence rate ratio (IRR) for all cancers | Cancer occurrence after a lag period (2 years)
  age and sex-standardized IRRs for all cancers for CT-exposed versus unexposed patients.

OTHER OUTCOMES:
Sensitivity analysis | Cancer occurrence after different lag periods (6 months, 1 year, 3 years and 5 years)
  Various lag periods will be applied for the outcomes.
Subgroup analysis by subsequent CT scans conducted more than 7 days after appendectomy | CT undergone more than 7 days after appendectomy will be counted.
  IRR in patients who underwent CT after appendectomy IRR in patients who did not undergo CT after appendectomy
Subgroup analysis | Cancer occurrence after a lag period (2 years)
  by age and sex

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bunadang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No